CLINICAL TRIAL: NCT04563000
Title: Impact of Vitamin C on Biomarkers of Neurologic Injury in Patients With Return of Spontaneous Circulation After Out-of-Hospital Cardiac Arrest
Brief Title: Impact of Vitamin C on Biomarkers of Neurologic Injury in Survivors of Cardiac Arrest
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VitC
Record Dates: First submitted 2020-09-10; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Heart Arrest, Out-Of-Hospital; Biomarkers; Oxidative Stress; Neurological Injury
Keywords: vitamin C; biomarkers; brain injury; cardiac arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Trauma, Nervous System; Brain Injuries; Heart Arrest | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): Group of patients that will receive vitamin C (ascorbic acid 1,5 g mixed with 0,9 % solution of sodium chloride 100 ml every 12 hours for 4 days intravenously).
  Interventions: Drug: Vitamin C
- Placebo (Placebo Comparator): Group of patients that will receive placebo (0,9 % solution of sodium chloride 100 ml every 12 hours for 4 days intravenously).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin C — Ascorbic acid 1,5 g intravenously every 12-hours for 4 consecutive days
  Arms: Vitamin C
Drug: Placebo — 0,9 % solution of sodium chloride 100 ml intravenously every 12-hours for 4 consecutive days
  Arms: Placebo

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) is one of the leading cause of death in the world. In Slovenia approximately 25% of resuscitated patients survives to discharge from hospitals, usually with poorer functional status.

One of key pathophysiological process responsible for poorer functional status is global hypoxic-ischemic injury, which is two-stage. Primary stage occurs immediately after cardiac arrest due to cessation of blood flow. With return of spontaneous circulation a secondary injury occurs, of which the leading process is an imbalance between oxygen delivery and consumption. Reperfusion exposes ischemic tissue to oxygen, resulting in the formation of large amounts of highly reactive oxygen species (ROS) within minutes. ROS lead to oxidative stress, which causes extensive damage to cell structures and leads to cell death. Consequently, necrosis and apoptosis are responsible for organ dysfunction and functional outcome of these patients.

Such injury of neural tissue causes brain damage, which is ultimately responsible for poor neurological and thus functional outcome of OHCA survivors. The extent of brain damage can be determined in several ways: clinically by assessing quantitative and qualitative consciousness and the presence of involuntary movements in an unconscious patient, by assessing activity on electroencephalographic record, by imaging of the brain with computed tomography and magnetic resonance imaging, as well as by assessing levels of biological markers of brain injury. Of the latter, the S-100b protein and neuron-specific enolase have been shown to be suitable for such assessment.

Oxidative stress is counteracted by the body with endogenous antioxidants that balance excess free radicals and stabilize cellular function. Vitamin C (ascorbic acid) is the body's main antioxidant and is primarily consumed during oxidative stress. Large amounts of ROS rapidly depletes the body's vitamin C stores.

Humans cannot synthesise vitamin C and enteral uptake of vitamin C is limited by transporter saturation. On the other hand, parenteral (venous) dosing of vitamin C can achieve concentrations of vitamin C above physiological and thus produce a stronger antioxidant effect. The beneficial effect of parenteral dosing of vitamin C has been establish in several preclinical and clinical studies in patients with ischemic stroke and cardiac arrest.

The investigators hypothesize that there is a similarly beneficial effect of vitamin C in survivors of OHCA.

ELIGIBILITY:
Inclusion Criteria:

- comatose survivors of out-of-hospital arrest

Exclusion Criteria:

* patients with trauma, asphyxia, drowning or electrocution as a cause of cardiac arrest
* history of oxalate nephropathy or nephrolithiasis, glucose-6-phosphate dehydrogenase deficiency, and hemochromatosis
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of neurological injury | 5th day
  Serum levels of protein S-100b and neuron-specific enolase.

SECONDARY OUTCOMES:
Brain imaging (CT and MRI) | 3rd-10th day
  Unconscious survivors will have first brain imaging on the 3rd day, if still unconscious, second imaging around the 10th day. Imaging results will be descriptive (normal or pathological with signs of global ischemic injury: generalised edema, reduced grey and white matter differentiation, obliteration of the sulci). Second image will be compared to the first.
Electroencephalography (EEG) | 3rd-10th day
  Unconscious survivors will have first EEG on the 3rd day, if still unconscious, second imaging around the 10th day. EEG results will be descriptive (normal or pathological with background suppression with or without periods of bursts, with or without response to external stimulus and similar patterns). Second EEG will be compared to the first.
Evaluation of pupils | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  Pupils size, reactivity and symmetry on admission and during hospitalisation will be observed daily.
Evaluation of involuntary movements | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  The presence of involuntary movements will be observed daily.
Evaluation of GCS | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  Level of consciousness will be determined daily with Glasgow Coma Scale (GCS).
Evaluation of FOUR | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  Level of consciousness will be determined daily with Full Outline of UnResponsiveness (FOUR) score.
Cerebral Performance Category | from admission till discharge from ICU or death (whatever comes first)
  Cerebral Performance Category (CPC) at discharge will be recorded.
Left ventricular ejection fraction | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  Left ventricular ejection fraction (first, last, best, worst), determined by ultrasound will be noted.
Arrhythmias | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  Presence of arrhythmias and the need for treating them will be recorded.
Evaluation of heart failure | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  Clinical evaluation of heart failure according to Killip-Kimball classification will be performed (worst result).
Serum troponin level | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  Serum troponin levels will be determined (on admission, minimal, maximal).
Serum Brain natriuretic peptide | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  Serum brain natriuretic peptide levels will be determined (on admission, minimal, maximal).
Vasopressor and/or inotrope need | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  The need for vasopressors and inotropes will be noted, along with the name of the substance, maximal dosage and duration.
Mechanical ventilation | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  Days and hours of mechanical ventilation will be noted.
Kidney failure | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  The need for renal replacement therapy (and consecutive day of such therapy) will be recorded.
Serum urea levels | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  Serum levels of urea will be recorded (on admission, minimal, maximal).
Serum creatinine levels | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  Serum creatinine levels will be recorded (on admission, minimal, maximal).
Serum C-reactive protein levels | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  Serum C-reactive protein levels will be determined (on admission, minimal, maximal).
Serum procalcitonin levels | from admission until 14 days or till discharge from ICU or death (whatever comes first)
  Serum procalcitonin levels will be determined (on admission, minimal, maximal).

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Markota, MD, PhD, Assist. Prof., Study Chair — University Medical Centre Maribor
Locations (1):
- University Medical Centre Maribor, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grasner JT, Lefering R, Koster RW, Masterson S, Bottiger BW, Herlitz J, Wnent J, Tjelmeland IB, Ortiz FR, Maurer H, Baubin M, Mols P, Hadzibegovic I, Ioannides M, Skulec R, Wissenberg M, Salo A, Hubert H, Nikolaou NI, Loczi G, Svavarsdottir H, Semeraro F, Wright PJ, Clarens C, Pijls R, Cebula G, Correia VG, Cimpoesu D, Raffay V, Trenkler S, Markota A, Stromsoe A, Burkart R, Perkins GD, Bossaert LL; EuReCa ONE Collaborators. EuReCa ONE-27 Nations, ONE Europe, ONE Registry: A prospective one month analysis of out-of-hospital cardiac arrest outcomes in 27 countries in Europe. Resuscitation. 2016 Aug;105:188-95. doi: 10.1016/j.resuscitation.2016.06.004. Epub 2016 Jun 16. PMID 27321577
- [Background] Nolan JP, Neumar RW, Adrie C, Aibiki M, Berg RA, Bottiger BW, Callaway C, Clark RS, Geocadin RG, Jauch EC, Kern KB, Laurent I, Longstreth WT, Merchant RM, Morley P, Morrison LJ, Nadkarni V, Peberdy MA, Rivers EP, Rodriguez-Nunez A, Sellke FW, Spaulding C, Sunde K, Hoek TV. Post-cardiac arrest syndrome: epidemiology, pathophysiology, treatment, and prognostication. A Scientific Statement from the International Liaison Committee on Resuscitation; the American Heart Association Emergency Cardiovascular Care Committee; the Council on Cardiovascular Surgery and Anesthesia; the Council on Cardiopulmonary, Perioperative, and Critical Care; the Council on Clinical Cardiology; the Council on Stroke. Resuscitation. 2008 Dec;79(3):350-79. doi: 10.1016/j.resuscitation.2008.09.017. Epub 2008 Oct 28. PMID 18963350
- [Background] Sekhon MS, Ainslie PN, Griesdale DE. Clinical pathophysiology of hypoxic ischemic brain injury after cardiac arrest: a "two-hit" model. Crit Care. 2017 Apr 13;21(1):90. doi: 10.1186/s13054-017-1670-9. PMID 28403909
- [Background] Wijdicks EF, Hijdra A, Young GB, Bassetti CL, Wiebe S; Quality Standards Subcommittee of the American Academy of Neurology. Practice parameter: prediction of outcome in comatose survivors after cardiopulmonary resuscitation (an evidence-based review) [RETIRED]: report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2006 Jul 25;67(2):203-10. doi: 10.1212/01.wnl.0000227183.21314.cd. PMID 16864809
- [Background] Calderon LM, Guyette FX, Doshi AA, Callaway CW, Rittenberger JC; Post Cardiac Arrest Service. Combining NSE and S100B with clinical examination findings to predict survival after resuscitation from cardiac arrest. Resuscitation. 2014 Aug;85(8):1025-9. doi: 10.1016/j.resuscitation.2014.04.020. Epub 2014 Apr 30. PMID 24795283
- [Background] Shinozaki K, Oda S, Sadahiro T, Nakamura M, Abe R, Nakada TA, Nomura F, Nakanishi K, Kitamura N, Hirasawa H. Serum S-100B is superior to neuron-specific enolase as an early prognostic biomarker for neurological outcome following cardiopulmonary resuscitation. Resuscitation. 2009 Aug;80(8):870-5. doi: 10.1016/j.resuscitation.2009.05.005. Epub 2009 Jun 17. PMID 19535196
- [Background] Spoelstra-de Man AME, Elbers PWG, Oudemans-van Straaten HM. Making sense of early high-dose intravenous vitamin C in ischemia/reperfusion injury. Crit Care. 2018 Mar 20;22(1):70. doi: 10.1186/s13054-018-1996-y. PMID 29558975
- [Background] Levine M, Padayatty SJ, Espey MG. Vitamin C: a concentration-function approach yields pharmacology and therapeutic discoveries. Adv Nutr. 2011 Mar;2(2):78-88. doi: 10.3945/an.110.000109. Epub 2011 Mar 10. PMID 22332036
- [Background] Tsai MS, Huang CH, Tsai CY, Chen HW, Lee HC, Cheng HJ, Hsu CY, Wang TD, Chang WT, Chen WJ. Ascorbic acid mitigates the myocardial injury after cardiac arrest and electrical shock. Intensive Care Med. 2011 Dec;37(12):2033-40. doi: 10.1007/s00134-011-2362-6. Epub 2011 Sep 28. PMID 21953354
- [Background] Tsai MS, Huang CH, Tsai CY, Chen HW, Cheng HJ, Hsu CY, Chang WT, Chen WJ. Combination of intravenous ascorbic acid administration and hypothermia after resuscitation improves myocardial function and survival in a ventricular fibrillation cardiac arrest model in the rat. Acad Emerg Med. 2014 Mar;21(3):257-65. doi: 10.1111/acem.12335. PMID 24628750
- [Background] Gao F, Yao CL, Gao E, Mo QZ, Yan WL, McLaughlin R, Lopez BL, Christopher TA, Ma XL. Enhancement of glutathione cardioprotection by ascorbic acid in myocardial reperfusion injury. J Pharmacol Exp Ther. 2002 May;301(2):543-50. doi: 10.1124/jpet.301.2.543. PMID 11961055
- [Background] Nishinaka Y, Sugiyama S, Yokota M, Saito H, Ozawa T. The effects of a high dose of ascorbate on ischemia-reperfusion-induced mitochondrial dysfunction in canine hearts. Heart Vessels. 1992;7(1):18-23. doi: 10.1007/BF01745863. PMID 1583008
- [Background] Basili S, Tanzilli G, Mangieri E, Raparelli V, Di Santo S, Pignatelli P, Violi F. Intravenous ascorbic acid infusion improves myocardial perfusion grade during elective percutaneous coronary intervention: relationship with oxidative stress markers. JACC Cardiovasc Interv. 2010 Feb;3(2):221-9. doi: 10.1016/j.jcin.2009.10.025. PMID 20170881
- [Background] Dingchao H, Zhiduan Q, Liye H, Xiaodong F. The protective effects of high-dose ascorbic acid on myocardium against reperfusion injury during and after cardiopulmonary bypass. Thorac Cardiovasc Surg. 1994 Oct;42(5):276-8. doi: 10.1055/s-2007-1016504. PMID 7863489
- [Background] Henry PT, Chandy MJ. Effect of ascorbic acid on infarct size in experimental focal cerebral ischaemia and reperfusion in a primate model. Acta Neurochir (Wien). 1998;140(9):977-80. doi: 10.1007/s007010050201. PMID 9842436
- [Background] Huang J, Agus DB, Winfree CJ, Kiss S, Mack WJ, McTaggart RA, Choudhri TF, Kim LJ, Mocco J, Pinsky DJ, Fox WD, Israel RJ, Boyd TA, Golde DW, Connolly ES Jr. Dehydroascorbic acid, a blood-brain barrier transportable form of vitamin C, mediates potent cerebroprotection in experimental stroke. Proc Natl Acad Sci U S A. 2001 Sep 25;98(20):11720-4. doi: 10.1073/pnas.171325998. PMID 11573006
- [Background] Lagowska-Lenard M, Stelmasiak Z, Bartosik-Psujek H. Influence of vitamin C on markers of oxidative stress in the earliest period of ischemic stroke. Pharmacol Rep. 2010 Jul-Aug;62(4):751-6. doi: 10.1016/s1734-1140(10)70334-0. PMID 20885017